CLINICAL TRIAL: NCT03726073
Title: Effect of Transcutaneous Acupoint Electrical Acupoint Stimulation Combined With Auricular Acupressure on Postoperative Delirium in Elderly Patients Undergoing Major Abdominal Surgery: a Pragmatic Randomized Clinical Trial
Brief Title: Acupoint Stimulation Improve Postoperative Delirium in Elderly Patients
Acronym: AICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, principle investigator, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJH-A-20181001
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Complications; Postoperative Delirium
Keywords: Delirium; Elderly patients; Transcutaneous acupoint electrical acupoint stimulation; Auricular acupressure
MeSH Terms: conditions — Postoperative Complications; Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: transcutaneous electrical acupoint stimulation and auricular acupressure is given by an investigator who is not involved in anesthesia and outcome assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Electrical stimulation will be given 30min before anesthesia and during surgery, auricular acupressure will be given in postoperative 3 days
  Interventions: Device: Transcutaneous acupoint electrical acupoint stimulation(TEAS) and auricular acupressure
- Non-intervention group (Sham Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Transcutaneous acupoint electrical acupoint stimulation(TEAS) and auricular acupressure — Bilaterally Hegu (LI4), Neiguan (PC6) and Zusanli (ST36) will be used as the TEAS acupoints. Six acupoints (Shenmen, Point Zero, subcortex, heart, liver, and endocrine) located on ears will be used as the auricular acupressure points.
  Arms: Intervention group
Other: Usual care — Patients in this group only receive usual care developed by the study hospital
  Arms: Non-intervention group

SUMMARY:
Postoperative delirium is with increased incidence in elderly patients. Previous studies have shown that acupuncture related techniques could induce protection against brain ischemia and improve outcome after cerebral diseases. In this study the effect of transcutaneous electrical acupoint stimulation combined with auricular acupressure on postoperative delirium will be evaluated.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is an acute neurological disorder that commonly happens between postoperative days 1 and 3 and more common reported in elderly patients. The rate of delirium differs depending on the patients' characteristics, surgery types and setting of health care. The prevalence of delirium range from 18% to 35 % in a general medical service, and up to half of older patients postoperatively. It has been documented that POD is associated with an increase in mortality and morbidity, increased use of hospital resources, and higher cost of health care. The conventional preventive methods for delirium have focused on minimization or elimination of the predisposing and precipitating factors. Yet, few effective therapies are available for treating POD. New treatments are needed to reduce the prevalence and severity of delirium.

Complementary therapies, particularly acupuncture, have gained increasing attention for their possible value in the prevention and treatment of neurological disorders. Both basic and clinical studies have suggested that acupuncture may be beneficial to postoperative delirium. In functional MRI studies of healthy subjects and nervous system dysfunction patients, acupuncture has been shown to stimulate hippocampus, amygdala and insula, areas of the brain associated with memory, cognition and emotion.

In the clinical, TEAS has been reported to be effective in alleviating delirium in elderly patients with silent lacunar infarction. Evidence also showed that auricular acupunctures are efficacious for preventing postoperative agitation in geriatric patients

Given evidences of the possible efficacy of TEAS and auricular acupressure, we aim to do a 2-arm, randomized, controlled, single-blinded, pragmatic trial to investigate whether transcutaneous electrical acupoint stimulation combined with auricular acupressure is more effective in reducing postoperative delirium in elderly patients than usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective abdominal surgery under general anesthesia
* American Society of Anesthesiologists (ASA) physical status class≤Ⅲ;
* Mini mental state examination (MMSE) score>20;

Exclusion Criteria:

* Implantation of a cardiac pacemaker, cardioverter, defibrillator or internal hearing aids;
* Documented alcohol or substance abuse within 3 months before surgery;
* Dermatological conditions or frail skin;
* Dysesthesia or infection over the acupoint stimulation skin area;
* Limb abnormalities;
* Allergy to ECG pads;
* Use of psychoactive medications;
* Severe visual or auditory impairment;
* Preoperative history of schizophrenia, epilepsy, parkinsonism, depression, or myasthenia gravis;
* Brain injury or neurosurgery.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | From the end of surgery to 7 days after surgery
  In postoperative 7 days or during patients stay in hospital if discharged within 7 days
The severity of delirium | From the end of surgery to 7 days after surgery or during patients stay in hospital if discharged within 7 days
  Assessed by memorial delirium assessment scale (MDAS)

SECONDARY OUTCOMES:
Postoperative pain | 24h, 48h, 72h after surgery
  Postoperative pain both at rest and with movement using Numeric Rating Scale (NRS)
S100B level | Before surgery and at the end of the surgery
  Serum
Neuron-specific enolase level | Before surgery and at the end of the surgery
  Serum
Brain-derived neurotrophic factor level | Before surgery and at the end of the surgery
  Serum
Tumor necrosis factor-α level | Before surgery and at the end of the surgery
  Serum
Interleukin- 6 level | Before surgery and at the end of the surgery
  Serum
Aquaporin-4 level | Before surgery and at the end of the surgery
  Serum
Postoperative sleep qualiy | 4 days after surgery
  Sleep quality within postoperative 4 days using Pittsburgh sleep quality index (PSQI)
Length of stay in hospital after sugery | From the day of suregry to discharge from surgery
  Days
Interleukin-10 level | Before surgery and at the end of the surgery
  Serum
Matrix metalloproteinase 9 level | Before surgery and at the end of the surgery
  Serum
Tau protain level | Before surgery and at the end of the surgery
  Serum
β-Amyloid1-42 level | Before surgery and at the end of the surgery
  Serum

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Lu, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be available for sharing after publishing, including data of the outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data of the study will be available for sharing after publishing on peer-reviewed journals, and will be available for 5 years

REFERENCES:
- [Background] Gao F, Zhang Q, Li Y, Tai Y, Xin X, Wang X, Wang Q. Transcutaneous electrical acupoint stimulation for prevention of postoperative delirium in geriatric patients with silent lacunar infarction: a preliminary study. Clin Interv Aging. 2018 Oct 24;13:2127-2134. doi: 10.2147/CIA.S183698. eCollection 2018. PMID 30425466
- [Background] Arai YC, Ito A, Hibino S, Niwa S, Ueda W. Auricular Acupunctures are Effective for the Prevention of Postoperative Agitation in Old Patients. Evid Based Complement Alternat Med. 2010 Sep;7(3):383-6. doi: 10.1093/ecam/nep172. Epub 2009 Oct 29. PMID 19875431
- [Background] Scholz AF, Oldroyd C, McCarthy K, Quinn TJ, Hewitt J. Systematic review and meta-analysis of risk factors for postoperative delirium among older patients undergoing gastrointestinal surgery. Br J Surg. 2016 Jan;103(2):e21-8. doi: 10.1002/bjs.10062. Epub 2015 Dec 16. PMID 26676760
- [Background] Matsumoto-Miyazaki J, Ushikoshi H, Miyata S, Miyazaki N, Nawa T, Okada H, Ojio S, Ogura S, Minatoguchi S. Acupuncture and Traditional Herbal Medicine Therapy Prevent Deliriumin Patients with Cardiovascular Disease in Intensive Care Units. Am J Chin Med. 2017;45(2):255-268. doi: 10.1142/S0192415X17500161. Epub 2017 Feb 23. PMID 28231740
- [Derived] Fan Q, Lei C, Wang Y, Yu N, Wang L, Fu J, Dong H, Lu Z, Xiong L. Transcutaneous Electrical Acupoint Stimulation Combined With Auricular Acupressure Reduces Postoperative Delirium Among Elderly Patients Following Major Abdominal Surgery: A Randomized Clinical Trial. Front Med (Lausanne). 2022 Jun 15;9:855296. doi: 10.3389/fmed.2022.855296. eCollection 2022. PMID 35783617